CLINICAL TRIAL: NCT03412630
Title: Perfusion CT to Predict Progression-Free Survival and Response Rate in Bevacizumab Treatment of Platinum-Resistant Persistent or Recurrent Epithelial Ovarian, Fallopian Tube, or Peritoneal Carcinoma
Brief Title: Perfusion CT in Predicting Outcomes in Ovarian, Fallopian, or Peritoneal Cancer With Bevacizumab
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor accrual
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EAE161; NCI-2017-01029 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAE161 (Other: ECOG-ACRIN Cancer Research Group); EAE161 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2018-01-22; First posted 2018-01-26 (Actual); Results first posted 2022-09-27 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Cytidine Triphosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Diagnostic (computed tomography perfusion imaging) (Experimental): Patients undergo computed tomography perfusion imaging at baseline and on day 15 after initiation of standard of care bevacizumab treatment and before the second dose.
  Interventions: Radiation: Computed Tomography Perfusion Imaging

INTERVENTIONS:
Radiation: Computed Tomography Perfusion Imaging — Undergo computed tomography perfusion imaging

SUMMARY:
This phase II trial studies how well computed tomography perfusion imaging works in predicting outcomes in patients with ovarian, fallopian tube, or primary peritoneal cancer who are receiving bevacizumab. Computed tomography perfusion imaging monitors the effects of the drug treatment on the blood flow to the tumor, and may help to predict whether a certain drug therapy is likely be successful in a patient with ovarian, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate whether those patients with an increase in perfusion computed tomography (CT) tumor blood flow (BF) from T0 to T1 demonstrate poorer progression-free survival (PFS) compared to those patients with a decrease in BF from T0 to T1, among platinum-resistant, recurrent ovarian cancer patients treated with bevacizumab.

SECONDARY OBJECTIVES:

I. To evaluate whether change in perfusion CT tumor BF from T0 to T1, as a continuous variable, is associated with PFS.

II. To evaluate whether changes in perfusion CT tumor blood volume (BV) or permeability surface product area (PS) from T0 to T1 are associated with PFS.

III. To evaluate whether changes in perfusion CT tumor BF, BV, or PS from T0 to T1 are associated with response rate according to the standard anatomic response evaluation criteria (RECIST 1.1).

IV. To identify which combination of perfusion CT parameters, including tumor BF, BV, and PS, can serve to optimally distinguish patients in terms of PFS outcome.

V. To evaluate whether the association between change in perfusion CT parameters and treatment outcome (PFS or tumor response) is stable when analyzed with various commercially-available post-processing software.

TERTIARY OBJECTIVES:

I. In the subset of patients with multiple, eligible perfusion target lesions within the CT imaging volume, describe the variability of perfusion CT changes across different lesions within the same patient, and evaluate the impact of multiple target lesions on the association between change in perfusion CT parameters and PFS.

II. In a subset of patients, measure the reliability of perfusion CT parameters by analyzing the same perfusion imaging dataset using different readers and different post-processing software.

OUTLINE:

Patients undergo computed tomography perfusion imaging at baseline and on day 15 after initiation of standard of care bevacizumab treatment and before the second dose.

After completion of study, patients are followed up every 8 weeks for up to 18 months.

ELIGIBILITY:
Inclusion Criteria:

* REGISTRATION TO STEP 0
* Patient must have epithelial ovarian, fallopian tube, or primary peritoneal cancer

  * Patients with non-epithelial tumors or tumors with low malignant potential are excluded
* Patient must have suspected platinum-resistant disease (disease progression =< 6 months of platinum therapy)
* Patient must be expected to undergo therapy with bevacizumab in combination with paclitaxel, pegylated liposomal doxorubicin (PLD), or topotecan at recommended standard of care doses if suspected recurrence is confirmed with imaging
* Patient must be able and willing to provide written informed consent
* Patient must have a life expectancy of >= 3 months
* Patient must have adequate bone marrow, coagulation, renal, and hepatic function
* Patient must demonstrate an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Patient must not have undergone therapy with any anti-VEGF drug within previous 6 months
* Patient must not have undergone major surgery or radiotherapy to the pelvis or abdomen within previous 4 weeks
* Patients must not have known contraindications to bevacizumab, including but not limited to abdominal fistula, gastrointestinal (GI) perforation, intra-abdominal abscess, thrombotic or hemorrhagic disorders, uncontrolled hypertension or active clinically significant cardiovascular disease, non-healing wound, ulcer, or bone fracture within previous 4 weeks
* Patient must not have untreated or symptomatic central nervous system (CNS) metastasis
* Patient must not have another active (within past 3 years) or concurrent malignancy
* Patient must not have contraindication to iodinated contrast
* REGISTRATION TO STEP 1
* Patient must be evaluable using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
* Patient must have perfusion CT target lesion (e.g., >= 1 cm in both the long and short axis, at least one half of the tumor appears enhancing and solid on a contrast-enhanced scan or has an attenuation of >= 10 Hounsfield unit [HU] on the unenhanced CT scan) on a contrast-enhanced conventional CT
* Conventional chest abdomen and pelvis CT images demonstrating recurrent tumor must be submitted within 21 days from acquisition to the American College of Radiology (ACR) Core Lab
* Eligibility of a perfusion CT target lesion must be confirmed by the ACR Core Lab prior to study enrollment and the T0 perfusion CT scan

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2020-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Lee, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Only 1 participant was accrued. To comply with HIPAA requirements no data will be shared.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was accrued on December 13, 2018.
Period: Overall Study
Arm/Group | Diagnostic (Computed Tomography Perfusion Imaging)
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 1 participant was accrued and available for analysis. This is insufficient for any meaningful statistical analysis and all results have been suppressed to comply with HIPAA
Arm/Group | Diagnostic (Computed Tomography Perfusion Imaging)
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: years] — Numbers not provided to comply with HIPAA Population: Numbers not provided to comply with HIPAA
Sex: Female, Male [Count of Participants; unit: Participants] — Not provided due to limited data Population: Numbers not provided to comply with HIPAA
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Numbers not provided to comply with HIPAA

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: The PFS of patients with increased tumor blood flow (BF) from T0 to T1 will be compared with that of patients with decreased tumor BF from T0 to T1. Kaplan-Meier survival curves will be generated, and a two-sided log-rank test will be used to compare PFS between the two groups.
Time Frame: Time to progression or death from the T1 scan, assessed up to 18 months
Population: Analysis not performed due to lack of data. Only 1 participant was accrued and available for analysis. This is insufficient for any meaningful statistical analysis and thus no analyses were performed. To comply with HIPAA requirements, all data and results for this participant been suppressed .
Arm/Group | Diagnostic (Computed Tomography Perfusion Imaging)
Number analyzed (Participants) | 0

2. Secondary Outcome: Objective Response Rate
Description: Will be assessed by Response Evaluation Criteria in Solid Tumors version 1.1.
Time Frame: Up to 18 months
Population: Analyses not performed due to lack of data. Only 1 participant was accrued and available for analysis. This is insufficient for any meaningful statistical analysis and thus no analyses were performed. To comply with HIPAA requirements, all data and results for this participant been suppressed .
Arm/Group | Diagnostic (Computed Tomography Perfusion Imaging)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were assessed at baseline imaging, and before second dose of Tx, up to 30 days..
Arm/Group | Diagnostic (Computed Tomography Perfusion Imaging)
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/30/NCT03412630/Prot_000.pdf
  • Informed Consent Form (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/30/NCT03412630/ICF_001.pdf